CLINICAL TRIAL: NCT01912196
Title: A Double-Blind, Placebo-Controlled, Randomized Add-On Study of MSI-195 (Methylation Sciences Inc. S-Adenosyl-L-Methionine, SAMe) For Patients With Major Depressive Disorder(MDD) Who Have Had An Inadequate Response to Current Antidepressant Therapy
Brief Title: Add-On Study of MSI-195 (S-Adenosyl-L-Methionine, SAMe) for Patients With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MSI Methylation Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSI-CP.002
Record Dates: First submitted 2013-07-26; First posted 2013-07-31 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSI-195 (Experimental): Patients randomized to the MSI-195 arm will receive treatment with 2 tablets (800 mg) of MSI-195 plus on-going antidepressant therapy (ADT).
  MSI-195 800 mg (two tablets) taken orally once a day in the morning on an empty stomach with water (food should be avoided for at least 1 hr after taking the study drug)
  Interventions: Drug: MSI-195
- Placebo (Placebo Comparator): Patients randomized to the placebo arm will receive 2 tablets placebo plus on-going antidepressant therapy (ADT).
  Placebo (two tablets) taken orally once a day in the morning on an empty stomach with water (food should be avoided for at least 1 hr after taking the study drug).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MSI-195
  Arms: MSI-195
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of 800 mg MSI-195 in reducing symptoms of depression in Major Depressive Disorder (MDD)patients with inadequate response to current antidepressant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Meets the Diagnostic and Statistical Manual of Mental Disorder, 4th Edition, Text Revision (DSM-IV-TR) criteria for Major Depressive Disorder (MDD)
* A total score of 16 or higher on the Hamilton Rating Scale for Depression- 17 item version (HAM-D17) at the Screening and Baseline Visits, with a score of ≥2 on mood item 1.
* Have experienced 1-4 prior Major Depressive Episodes. Patients with more than 5 lifetime episodes (including current episode) will require discussion with the medical monitor prior to inclusion.
* Failed 1-3 treatment regimens in the current depressive episode
* Received an adequate dose and duration of Antidepressant Therapy (ADT) (on ADT for at least 6 weeks with a stable dose for at least 3 weeks)

Exclusion Criteria:

* Failed 4 or more adequate treatment regimens in current episode of depression
* patient may have a significant risk for suicidal behavior during the course of their participation in the study
* Intolerance to SAMe; Prior use of MSI-195
* History of any of the following psychiatric disorders: eating disorder within 6 months; obsessive compulsive disorder, psychotic disorder, bipolar disorder, mental retardation, dementia or other forms of cognitive impairment at any time or alcohol or substance abuse
* >3X upper limit of normal (ULN) Alkaline Phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT); >1.5X ULN total bilirubin
* Pregnant or lactating women
* Any history of seizures, excluding febrile seizures
* Known positivity for human immunodeficiency virus

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in the total Hamilton Depression Rating Scale (HAM-D17) between randomization and end of study. | assessed from baseline to week 8 (end of study)
  Based on historical data, the standard deviation is assumed to range between 9 and 12. With a standard effect size of 0.367 a total of at least 120 evaluable patients per group are needed to provide 80% power with a two-sided 5% significance level. HAM-D17 will be derived from the Combined HAM-D28-MADRS Instrument.

SECONDARY OUTCOMES:
change in the total score of the Montgomery-Asberg Depression Rating Scale (MADRS) | collected at baseline, weeks 2, 4, 6, 7 and 8 (end of study)
  for the MADRS, the number and proportion of patients who are responders at the end of the study and the number and proportion of patients who are in remission at the end of the study will be summarized by treatment group, along with the difference and 95% confidence interval for the difference (based on the Wilson Score method).
change in total score of the Clinical Global Impression Improvement Scale (CGI-S) | assessed from baseline, weeks 2, 4, 7 and 8 (end of study)
  the number and proportion of patients who are responders at the end of the study and the number and proportion of patients who are in remission at the end of the study will be summarized by treatment group, along with the difference and 95% confidence interval for the difference (based on the Wilson Score method). Remission is defined as a score of 1 or 2.
change from randomization to each study visit in the total score of the Inventory of Depressive Symptomatology-Self Rated (IDS-SR30) | assessed on baseline visit, Week 2, 4, 6, and 8 (end of study).
  A response is defined as a reduction in the IDS-SR30 score of ≥50% and remission is defined as a score of ≤14.
Adverse events | collected at baseline, weeks 1, 2, 3, 4, 6, 8 and 9 (follow up)
  collected from signing informed consent through 7 days after the last dose of study treatment. Ascertained by qualified clinician.
Columbia Suicide Severity Rating Scale (C-SSRS) | assessed at baseline, weeks 2, 4, 6 and 8 (end of study)
  administered by qualified clinician

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - MSI Investigational Site, Birmingham, Alabama
  - MSI Investigational Site, Encino, California
  - MSI Investigational Site, Escondido, California
  - MSI Investigational Site, Garden Grove, California
  - MSI Investigational Site, Los Alamitos, California
  - MSI Investigational Site, Los Angeles, California
  - MSI Investigational Site, National City, California
  - MSI Investigational Site, Newport Beach, California
  - MSI Investigational Site, Oakland, California
  - MSI Investigational Site, Oceanside, California
  - MSI Investigational Site, Torrance, California
  - MSI Investigational Site, Jacksonville, Florida
  - MSI INvestigational Site, Kissimmee, Florida
  - MSI Investigational Site, Lauderhill, Florida
  - MSI Investigational Site, Orlando, Florida
  - MSI Investigational Site, Atlanta, Georgia
  - MSI Investigational Site, Hoffman Estates, Illinois
  - MSI Investigational Site, Towson, Maryland
  - MSI Investigational Site, Flowood, Mississippi
  - MSI Investigational Site, Las Vegas, Nevada
  - MSI Investigational Site, Marlton, New Jersey
  - MSI Investigational Site, Albuquerque, New Mexico
  - MSI Investigational Site, New York, New York
  - MSI Investigational Site, Rochester, New York
  - MSI Investigational Site, Canton, Ohio
  - MSI Investigational Site, Dayton, Ohio
  - MSI Investigational Site, Portland, Oregon
  - MSI Investigational Site, Memphis, Tennessee
  - MSI Investigational Site, Austin, Texas
  - MSI Investigational Site, Dallas, Texas
  - MSI Investigational Site, Houston, Texas
  - MSI Investigational Site, Murray, Utah
  - MSI Investigational Site, Bellevue, Washington

REFERENCES:
- [Derived] Targum SD, Cameron BR, Ferreira L, MacDonald ID. An augmentation study of MSI-195 (S-adenosylmethionine) in Major Depressive Disorder. J Psychiatr Res. 2018 Dec;107:86-96. doi: 10.1016/j.jpsychires.2018.10.010. Epub 2018 Oct 18. PMID 30368163